CLINICAL TRIAL: NCT05810753
Title: SPOONful: a Structured Prescription Of Oral Nutritional Supplementation for Community-dwelling Older Adults - a Feasibility Study
Brief Title: Oral Nutritional Supplementation and Community-dwelling Older Adults: a Feasibility Study
Acronym: SPOONful
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University of Leeds (Other); Aston University (Other); Food4Years Ageing Network (Unknown)
Responsible Party: Principal Investigator, Chris McLeod, Lecturer, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPOONful_13002
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Malnutrition; Healthy Aging
Keywords: Oral nutritional supplementation; Older adults; Prescription
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPOONful (Experimental): Participants will be asked to consume one ONS with their breakfast, and one with their lunch, daily for three weeks.
  Interventions: Behavioral: SPOONful
- Control (No Intervention): Participants will be asked to consume two ONS daily, in addition to their regular diet, for three weeks without any precise instruction regarding when to consume the ONS during the day (standard care).

INTERVENTIONS:
Behavioral: SPOONful — Participants will be asked to consume two ONS daily, in addition to their regular diet, for three weeks. Participants will be asked to consume one ONS with their breakfast, and one with lunch.
  Arms: SPOONful

SUMMARY:
The goal of this study is to assess the feasibility and acceptability to community-dwelling older adults of implementing a precise prescription of oral nutritional supplementation (the SPOONful intervention).

DETAILED DESCRIPTION:
Oral nutritional supplementation (ONS) can treat and prevent malnutrition in older adults (aged ≥70 years). However, older adults' adherence to ONS is poor (~ 37%). One specific influence that may impact adherence is how effectively ONS prescription corresponds with older-adults' typical daily eating patterns (i.e., eating three meals daily and snacking infrequently). Currently, prescription instructions for ONS provided by the UK's National Health Service/National Institute for Health and Care Excellent lack precision within daily eating patterns and place the onus on healthcare practitioners to determine effective implementation. Poor ONS adherence could be caused, in part, by this imprecise prescription.

This hypothesis is founded on research demonstrating the importance of behavioural habit strength in promoting health-behaviour engagement/maintenance. Medical research suggests that forming medication-taking routines/habits through 'piggybacking' (combining a new behaviour with an existing habit/routine) can improve long-term adherence by reducing novel, deliberative behaviours requiring additional cognitive and self-regulatory resources - this is particularly salient for older adults where cognitive decline is widely experienced and a clear barrier to engaging in novel behaviours. Piggybacking with medical care is a key, under explored and relevant direction of enquiry to improve ONS adherence.To explore the idea that a more precise prescription may increase adherence to ONS, a feasibility and acceptability study will be undertaken to provide an initial evaluation of the SPOONful intervention.

Consent will be sought from community-dwelling older adults who will be asked to take part in a two-day familiarisation phase to ensure they understand the protocol and do not dislike or have an adverse reaction to the ONS. They will then be randomised into the intervention or control group. In the intervention group, participants will be asked to consume two ONS at particular times of day for three weeks. In the control group, participants will engage in usual care for ONS, i.e., they will be asked to consume two ONS daily but without specific instruction as to when this should be. All participants will subsequently engage in a follow-up phase comprising interviews with participants. Participants will complete all phases at home. The data gathered will be used to inform the feasibility and acceptability of a later trial.

ELIGIBILITY:
Inclusion Criteria:

* Be aged ≥70 years.
* Be living independently in the community.
* Be able to self-feed.
* Score >12 on The Montreal Cognitive Assessment (5-minute telephone version).
* Not be classified as High Risk of Malnutrition as assessed by the Malnutrition Universal Screening Tool
* Not have a BMI ≥40.
* Not have diabetes, a diagnosed eating disorder, a history of gastric/digestive/metabolic/cardiovascular/anosmia/renal disease, galactosaemia or another issue negatively impacting eating.
* Not have an allergy/intolerance/dislike or previous experience of regularly taking ONS.
* Regularly eat breakfast and lunch (≥5 times per week).

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Attrition rate | From randomisation (post-familiarisation) to end of intervention week 3.
  The primary outcome is the feasibility and acceptability of the SPOONful intervention which includes an assessment of attrition rate which will be derived by dividing the number of withdrawn participants (calculated as the number of people retained to the end of the intervention/control period subtracted from the total number randomised) by the number originally randomised.
Completion of self-report data-collection booklet denoting ONS consumption | From start of week 1 to end of week 3
  The primary outcome is the feasibility and acceptability of the SPOONful intervention which includes an assessment of participants' ability to complete the self-report data-collection booklet denoting their ONS consumption. Completion of data-collection booklet with times of ONS intake will be calculated as the percentage of blank/incomplete data cells.
Daily consumption of Oral Nutritional Supplementation as per prescription. | From start of week 1 to end of week 3
  The primary outcome is the feasibility and acceptability of the SPOONful intervention which includes an assessment of daily consumption of ONS as prescribed will be measured as the percentage of instances where participants did not adhere to the prescription.

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Available upon request once the study findings have been published.
Supporting Information: Study Protocol, ICF
Time Frame: Intention to publish date 1/12/2024
Access Criteria: Anonymous data will be shared with all who request access via email for novel analyses or re-analysis of the study outcomes. This will be administered by Dr Chris McLeod.